CLINICAL TRIAL: NCT02772380
Title: Acute Extravascular Defibrillation Study
Brief Title: Acute Study to Collect Electrical Signals From the Heart Using a Special Lead
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Device Feasibility
Other Study IDs: ASD2; U1111-1179-2213 (Other: WHO)
Record Dates: First submitted 2016-04-27; First posted 2016-05-13 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-03

CONDITIONS: Tachycardia; Ventricular Arrhythmias
MeSH Terms: conditions — Tachycardia

STUDY DESIGN:
Intervention Model Description: Subjects who are undergoing a standard of care procedure will also undergo the ASD2 research procedure involving placing an investigational lead in the substernal space to gather electrograms during induced ventricular arrhythmias for future research/development.
Oversight: Data Monitoring Committee: No

ARMS (1):
- VT/ VF induction and defibrillation (Experimental): Ventricular Tachycardia and Ventricular Fibrillation (VT/VF) induction and termination through use of a defibrillator, will be carried out as the intervention in all subjects undergoing study procedures.
  Interventions: Device: Defibrillation following induction of VT/VF

INTERVENTIONS:
Device: Defibrillation following induction of VT/VF — Up to 10 attempts to induce two VF/VT episodes for defibrillation testing

SUMMARY:
The main purpose of this clinical study is to collect electrograms from an investigational lead placed in an extravascular space, for development of a future Implantable Cardioverter Defibrillator (ICD) system.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be undergoing surgical procedure for approved indications for:

  * cardiothoracic surgery where a midline sternotomy is planned, or
  * cardiothoracic surgery where a subxiphoid/paraxiphoid cut for a chest tube is planned, or
  * VT ablation procedure with epicardial access, or
  * implant of a subcutaneous ICD (S-ICD®), or implant of a transvenous ICD (single or dual chamber)
* Subject must be willing to provide Informed Consent
* Subject must be ≥ 18 years old

Exclusion Criteria:

* Subject has known hiatus hernia or moderate or worse pectus excavatum
* Subject had previous pericarditis or prior sternotomy
* Subject has known significant Right Ventricle/ Right Ventricular dilation
* Subject has hypertrophic cardiomyopathy
* Subject is pacemaker dependent
* Subject has known skin irritations due to the Covidien Multi-function defibrillation electrode
* Subject is considered to be at high risk for infection(1)
* Subject has Left Ventricular Ejection Fraction < 20% (most recent available LVEF measurement in the last 6 months)
* Subject has New York Heart Association Class IV
* Subject has myocardial infarction within the last 6 weeks
* Subject currently has unstable angina
* Subject has severe aortic stenosis
* Subject at high risk of stroke (2)
* Subject has Chronic Obstructive Pulmonary Disease and is oxygen dependent
* Subject has permanent AF and will not be adequately anticoagulated during the ASD2 Acute Testing procedure (3)
* Subject with an implanted active cardiac or non-cardiac device during the ASD2 Acute Testing procedure (e.g., ICD, S-ICD®, Pacemaker, Neuro stimulator)
* Subject is enrolled in a concurrent study that may confound the results of this study, without documented pre-approval from a Medtronic study manager
* Subject has any medical condition that would limit study participation
* Subject is pregnant, or of childbearing potential and not on a reliable form of birth control. Women of childbearing potential are required to have a negative pregnancy test within 7 days prior to the ASD2 Acute Testing procedure
* Subject meets exclusion criteria required by local law (e.g. age, breast feeding,etc.)
* Subject is legally incompetent

  1. Screening subjects at high risk for infection will be based on the local investigator judgment decision.
  2. Subjects who are at high risk for stroke should be screened according to local country guidelines or, in case of their absence, according to ACC/AHA/ESC 2006 Guidelines for High Risk Factors for Stroke (i.e. exclusion of subjects with previous stroke, TIA, or embolism; Mitral stenosis; prosthetic heart valve).
  3. Screening will be based on the local investigator judgment decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2016-05; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Number of extravascular electrograms collected during ventricular fibrillation or ventricular tachycardia episodes | Day of procedure
  Collect extravascular EGMs during induced VF/VT and intrinsic rhythms directly from an investigational lead placed in the extravascular space to be used for development of a future ICD.

CONTACTS AND LOCATIONS:
Locations (36):
- United States (14):
  - Arizona Arrhythmia Consultants, Scottsdale, Arizona
  - Hartford Hospital, Hartford, Connecticut
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Iowa Heart Center, Des Moines, Iowa
  - University of Maryland Medical Center, Baltimore, Maryland
  - Mayo Clinic (Rochester MN), Rochester, Minnesota
  - Lourdes Cardiology Services, Cherry Hill, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - New York-Presbytarian Hospital / Well Cornell Medical Center, New York, New York
  - NYU Langone Medical Center, New York, New York
  - Raleigh Cardiology Associates, Raleigh, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Lancaster General Hospital, Lancaster, Pennsylvania
- Austin Hospital, Heidelberg, Victoria, Australia
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - UZ Leuven - Campus Gasthuisberg, Leuven
- Canada (3):
  - Royal Columbian Hospital, New Westminster, British Columbia
  - London Health Sciences Centre - University Campus, London, Ontario
  - Institut Universitaire de Cardiologie et de Pneumologie de Québec (IUCPQ), Québec, Quebec
- Prince of Wales Hospital, Kowloon, Hong Kong
- Semmelweis University, Budapest, Hungary
- Netherlands (3):
  - Academisch Medisch Centrum (AMC), Amsterdam
  - Maastricht Universitair Medisch Centrum, Maastricht
  - St. Antonius Ziekenhuis, Nieuwegein
- Christchurch Hospital, Christchurch, New Zealand
- Poland (2):
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow
  - Slaskie Centrum Chorob Serca, Zabrze
- Hospital Universitario Reina Sofia, Córdoba, Spain
- Taiwan (3):
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (4):
  - Liverpool Heart and Chest Hospital, Liverpool
  - King's College of London, London
  - John Radcliffe Hospital Oxford, Oxford
  - Southampton General Hospital - University Hospital Southampton NHS Foundation Trust, Southampton